CLINICAL TRIAL: NCT01572337
Title: Reducing the Need for Intensive Care Unit in Hospitalized Patients With Early Respiratory Failure Using the Non-invasive Ventilation Technique. A Multicentre Randomized Study.
Brief Title: Early Non-invasive Ventilation Outside the Intensive Care Unit
Acronym: NAVIGATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Head of Research, Department of Anesthesiology and Intensive Care, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VP/96/ER/mm
Record Dates: First submitted 2012-03-16; First posted 2012-04-06 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Early Acute Respiratory Failure
Keywords: NIV; acute respiratory failure; hypoxia; hypercapnia; non-invasive ventilation; hospital ward
MeSH Terms: conditions — Hypoxia; Hypercapnia | interventions — Noninvasive Ventilation; Standard of Care

ARMS (2):
- NIV (Experimental): Non-invasive ventilation
  Interventions: Procedure: Non-invasive ventilation
- Best available treatment (Other)
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Non-invasive ventilation — Early non-invasive ventilation will be given to patients at an early stage of acute respiratory failure
  Other Names: Noninvasive ventilation; NIV
  Arms: NIV
Other: Standard care
  Arms: Best available treatment

SUMMARY:
A large multicentre, randomized, controlled trial to demonstrate that non invasive ventilation given at an early stage of acute respiratory failure (ARF) outside the intensive care unit (ICU) can prevent the deterioration of ARF and the need for ICU when compared to the best available treatment usually performed in the non-ICU wards.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age >= 18 years
* Admission in a non-intensive-care department
* Radiological evidence of new pulmonary consolidation or atelectasis
* Peripheral Oxygen saturation less than 92% while breathing room air or PaO2/FiO2 ratio less than 300 at blood gas analysis
* Decompensated hypercapnia (pCO2 > 45 mmHg and pH < 7.35)
* Clinical signs of respiratory distress (dyspnoea, utilization of accessory respiratory muscles, paradox movements of thoraco-abdominal wall) in air.

Exclusion Criteria:

* Respiratory failure due to chronic obstructive pulmonary disease exacerbation, defined as PaCO2 > 45 and pH < 7.35 (in these patients NIV is considered to be the standard/first line treatment and we do not want to deny these patients the opportunity to receive this treatment because of randomization)
* Severe, hypercapnic ARF defined as PaCO2 > 45 and pH < 7.30
* Severe, hypoxic ARF defined as PaO2/FiO2 < 200
* Need for immediate mechanical ventilation or ICU as judged by the ICU physician in charge
* Extremely poor short term prognosis (imminent death with decision for palliative treatment only)
* Invasive or non-invasive mechanical ventilation during the same hospitalization due to respiratory failure.
* Clear contraindication to NIV treatment: respiratory arrest, failure to correct positioning of a face mask, hemodynamic instability due to hypotensive shock, ongoing myocardial ischemia, arrhythmia, massive bleeding from upper gastrointestinal tract, patient uncooperative and upset, inability to protect airways, alterations of deglutition, inability to clear secretion also with external aspiration, multiple organs dysfunction, recent surgery of airways or upper gastrointestinal tract, not-drained pneumothorax, bowel obstruction, active vomit.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Number of patients who will need admission to the Intensive Care Unit care for severe acute respiratory failure | participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (14):
- University of Thessaly, Larissa, Greece
- Italy (12):
  - Ospedale San Raffaele di Milano, Milan, MI
  - Ospedale Cesare Arrigo, Alessandria, Piedmont
  - Ospedale di Novara, Novara, Piedmont
  - Ospedale Civile di Asti, Asti
  - Spedali Civili, Brescia
  - Asl 3 Genovese, Genova
  - Ospedali Galliera, Genova
  - AOU Pisana, Pisa
  - Grande Ospedale Metropolitano, Reggio Calabria
  - Aurelia Hospital, Roma
  - Policlinico A. Gemelli, Roma
  - Azienda Ospedaliera San Giovanni Battista Molinette, Torino
- Astana Medical University, Kazakhstan, Kazakhstan

REFERENCES:
- [Background] Cabrini L, Nobile L, Plumari VP, Landoni G, Borghi G, Mucchetti M, Zangrillo A. Intraoperative prophylactic and therapeutic non-invasive ventilation: a systematic review. Br J Anaesth. 2014 Apr;112(4):638-47. doi: 10.1093/bja/aet465. Epub 2014 Jan 19. PMID 24444661
- [Background] Cabrini L, Plumari VP, Nobile L, Olper L, Pasin L, Bocchino S, Landoni G, Beretta L, Zangrillo A. Non-invasive ventilation in cardiac surgery: a concise review. Heart Lung Vessel. 2013;5(3):137-41. PMID 24364004
- [Result] Monti G, Cabrini L, Kotani Y, Brusasco C, Kadralinova A, Giardina G, Chalkias A, Nakhnoukh C, Pantazopoulos I, Oliva FM, Dazzi F, Roasio A, Baiardo Redaelli M, Tripodi VF, Cucciolini G, Belletti A, Vaschetto R, Maj G, Borghi G, Savelli F, Boni S, D'Amico F, Cavallero S, Labanca R, Tresoldi M, Marmiere M, Marzaroli M, Moizo E, Monaco F, Nardelli P, Pieri M, Plumari V, Scandroglio AM, Turi S, Corradi F, Konkayev A, Landoni G, Bellomo R, Zangrillo A; NAVIGATE Study Group. Early noninvasive ventilation in general wards for acute respiratory failure: an international, multicentre, open-label, randomised trial. Br J Anaesth. 2025 Feb;134(2):382-391. doi: 10.1016/j.bja.2024.11.023. Epub 2025 Jan 2. PMID 39753402
- [Derived] Cabrini L, Brusasco C, Roasio A, Corradi F, Nardelli P, Filippini M, Cotticelli V, Belletti A, Ferrera L, Antonucci E, Baiardo Redaelli M, Lattuada M, Colombo S, Olper L, Ponzetta G, Ananiadou S, Monti G, Severi L, Maj G, Giardina G, Biondi-Zoccai G, Benedetto U, Gemma M, Cavallero SSM, Hajjar LA, Zangrillo A, Bellomo R, Landoni G. Non-invAsive VentIlation for early General wArd respiraTory failurE (NAVIGATE): A multicenter randomized controlled study. Protocol and statistical analysis plan. Contemp Clin Trials. 2019 Mar;78:126-132. doi: 10.1016/j.cct.2019.02.001. Epub 2019 Feb 7. PMID 30739002